CLINICAL TRIAL: NCT00020202
Title: Phase II Study of FR901228 in Patients With Refractory or Progressive Small Cell or Non-Small Cell Lung Cancer
Brief Title: FR901228 in Treating Patients With Refractory or Progressive Small Cell Lung Cancer or Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068031; NCI-00-C-0123; NCI-1053; NCT00005656 (obsolete NCT alias)
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Recurrent Small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer
Keywords: adult solid tumor; body system/site cancer; cancer; extensive stage small cell lung cancer; genetic condition; lung cancer; non-small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; small cell lung cancer; solid tumor; stage III non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; stage, non-small cell lung cancer; stage, small cell lung cancer; thorax/respiratory cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Neoplasms; Genetic Diseases, Inborn; Lung Neoplasms | interventions — romidepsin

INTERVENTIONS:
Drug: FR901228

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of FR901228 in treating patients who have refractory or progressive small cell lung cancer or non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response of patients with refractory or progressive small cell or non-small cell lung cancer to FR901228.

II. Determine the ability of FR901228 to mediate apoptosis and target gene induction relative to tumor histology in these patients.

III. Determine the toxicity of this treatment in these patients.

PROTOCOL OUTLINE: Patients are stratified according to disease histology (small cell lung cancer vs non-small cell lung cancer).

Patients receive FR901228 IV over 4 hours on days 1 and 7. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL:

A total of 18-43 patients (9-21 per arm) will be accrued for this study within 18 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically or cytologically confirmed primary extensive stage small cell or unresectable non-small cell lung cancer Must have received or refused prior platinum-based chemotherapy and exhibited refractory or progressive disease Tumor must be accessible to biopsy by bronchoscopic or percutaneous fine needle aspiration technique Measurable disease outside of irradiated field or documented progression since irradiation Extrathoracic metastases allowed No active intracranial or leptomeningeal metastases Prior surgical resection or radiotherapy for intracranial metastatic disease allowed if: No evidence of active disease on 2 MRI scans AND No requirement for anticonvulsant medications or steroids to control residual symptoms --Prior/Concurrent Therapy-- Biologic therapy: At least 30 days since prior biologic therapy and recovered Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy, including nitrosoureas or mitomycin, and recovered No prior FR901228 No prior doxorubicin of total dose greater than 450 mg/m2 Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 30 days since prior radiotherapy and recovered At least 4 weeks since prior radiotherapy to the lung or mediastinum Surgery: See Disease Characteristics --Patient Characteristics-- Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Absolute neutrophil count at least 1,500/mm3 Hepatic: PT/PTT normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: Ejection fraction greater than 40% No unstable angina, congestive heart failure, or uncontrolled cardiac dysrhythmia No deep vein thrombosis requiring anticoagulation Pulmonary: No pulmonary embolism within past 6 months FEV1 and DLCO greater than 30% predicted pCO2 less than 50 mm Hg on room air pO2 greater than 60 mm Hg on room air Other: HIV negative No active infections Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schrump, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States